CLINICAL TRIAL: NCT04504942
Title: Basket Study of Leronlimab (PRO 140) in Patients With CCR5+ Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD09_Basket
Record Dates: First submitted 2020-06-10; First posted 2020-08-07 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — leronlimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leronlimab 525mg (Experimental): Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Interventions: Drug: Leronlimab

INTERVENTIONS:
Drug: Leronlimab — Drug: Leronlimab 525mg
  Other Names: Standard-of-care chemotherapy or radiotherapy

SUMMARY:
A single arm phase II study with 30 patients of leronlimab (PRO 140) in patients with CCR5+ locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Leronlimab (PRO 140) will be administered subcutaneously as weekly dose of 525 mg until disease progression or intolerable toxicity. Subjects participating in this study will be allowed to receive/continue standard-of-care chemotherapy or radiotherapy as per the dosing schedule included on the package insert.

In this study, patients will be evaluated for tumor response approximately every 3 months or according to institution's standard practice by CT, PET/CT or MRI with contrast (per treating investigator's discretion) using the same method as at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors:

   1. who have disease progression on standard therapy,
   2. who are receiving a standard anticancer treatment but no subsequent approved treatment would be available upon progression,
   3. who are unable to receive standard therapy, or
   4. for whom standard therapy does not exist.
2. Demonstrate CCR5 + by IHC (>10% of primary or metastatic tumor cells shows membranous staining and/or high predominance of CCR5+ tumor-infiltrating leukocytes completed at the reference laboratory of Dr. Hallgeir Rui at Medical College of Wisconsin).

   Note: This test will be done as part of the pre-screening period. It will be performed in archival metastatic tissue. If archival tissue is not available then, fresh biopsy will be done;
3. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (in case archival tissue is not available);
4. Patients must have measurable disease based on RECIST v1.1;
5. ≥ 18 years of age;
6. Patients must exhibit a/an ECOG performance status of 0-1;
7. Life expectancy of at least 6 months;
8. Patients must have adequate organ and bone marrow function within 28 days prior to registration, as defined below:

   * leukocytes ≥ 3,000/mcL;
   * absolute neutrophil count ≥ 1,500/mcL;
   * platelets ≥ 100,000/mcL;
   * total bilirubin: within normal institutional limits;
   * AST(SGOT) and ALT(SPGT) ≤ 2.5 X institutional upper limit of normal (ULN) (applicable to all patients, irrespective of liver disease or metastasis); and
   * creatinine: within normal institutional limits.
9. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
10. Females of child-bearing potential (FOCBP) and males must agree to use two medically accepted methods of contraception with hormonal or barrier method of birth control, or abstinence, prior to study entry, for the duration of study participation and for 60 days after the last dose of study drug (Refer to Appendix 1). Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; and
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months).
11. FOCBP must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
12. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days prior to enrollment;
2. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible;
3. Patients who have had prior exposure to CCR5 antagonists are not eligible;
4. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
5. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator;
6. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial; and
7. Is pregnant or breastfeeding, or expecting to conceive or have children within the projected duration of the trial, starting with the pre-screening or screening visit through the duration of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Study Director — CytoDyn, Inc.
Locations (1):
- Quest Clinical Research, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Leronlimab 525mg
Started | 16
Completed | 6
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — 7 patients were on-going at the time when study was closed by sponsor. | 7
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of leronlimab (PRO 140) were included in the baseline analysis population.
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Population: No birthday information was included for 1 patient.
  Participants
    number analyzed (Participants) | 15
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: No birthday information was included for 1 patient.
  years
    number analyzed (Participants) | 15
    (all) | 54.87 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), and Serious Adverse Events (SAEs).
Description: Adverse events were elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the investigator believed were clinically significant to the research subject were reported as adverse events.
Time Frame: From the time of first treatment (T1) until the last study visits completion (up to approximately 16 months)
Population: The population (N=16) consists of all subjects who received at least one dose of leronlimab (PRO 140).
Measure: Count of Participants; unit: Participants
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
Participants
  Adverse Events | 11
  Serious Adverse Events | 3

2. Primary Outcome: Changes in Eastern Cooperative Oncology Group (ECOG) Performance Status From Baseline to Subsequent Scheduled Visits
Description: The ECOG was utilized to assess the ability of patients to tolerate treatment. The ECOG is a 5-point scale, where a higher score indicates a greater lack of tolerance of the treatment. Response choices included: 0 = Asymptomatic; Fully active, able to carry on all pre-disease performance without restriction, 1 = Symptomatic but completely ambulatory; Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Symptomatic, <50% in bed during the day; Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours, 3 = Symptomatic, >50% in bed during the day; Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours, 4 = Bedbound; Completely disabled; cannot carry on any selfcare; totally confined to bed or chair, 5 = Dead.
Time Frame: From the time of first treatment (T1) until the last study visits completion (up to approximately 16 months)
Population: The population (N=16) consists of all subjects who received at least one dose of leronlimab (PRO 140). Subjects who had undefined change from baseline due to missing data were excluded from the analysis population.
Measure: Number; unit: Participants
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
Participants
  Participants with improved ECOG score | 2
  Participants with stable ECOG score | 2
  Participants with worsened ECOG score | 2
  Missing data | 10

3. Secondary Outcome: Progression Free Survival (PFS) Defined as Time in Months From the Date of First Study Treatment to the Date of Disease Progression or Death From Any Cause, Whichever Comes First.
Description: The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria was used for objective tumor response assessment (when disease is measurable and non- measurable); PFS is calculated from the date of first dose of leronlimab until date of clinical progressions.
Time Frame: The time in months from start of treatment to progression or death will be measured for all patients who receive at least one dose of study drug. Participants were followed on study until last study visit completion up to approximately 16 months.
Population: The population (N=16) consists of all subjects who received at least one dose of leronlimab (PRO 140). Censor subjects are all subjects who did not have a disease progression or death.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
months | 4.05 (2.758)

4. Secondary Outcome: Overall Response Rate (ORR, Defined as CR (Complete Response) + PR (Partial Response)) in Subjects With CCR5+ Locally Advanced or Metastatic Solid Tumors Treated With Leronlimab.
Description: Overall response rate is defined as the percentage of patients who achieve an overall response of complete response or partial response in the total number of evaluable patients, assessed by RECIST v1.1.
Time Frame: as for outcome 3
Population: The population consists of all subjects who received at least one dose of leronlimab (PRO 140). Subjects who had undefined change from baseline due to missing data were excluded from the analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 11
percentage of participants | 18.2

5. Secondary Outcome: Mean Time to New Metastases (TTNM)
Description: Recorded time from baseline metastatic disease (at time of enrollment) to the time of development of new metastasis in different site. New metastases in same site will be also recorded. TTNM will be calculated according to the formula: TTNM=(Date of new metastases - Date of first treatment) + 1.
Time Frame: From the time of first treatment (T1) until the last study visits completion (up to approximately 16 months).
Population: The population consists of all subjects who received at least one dose of leronlimab (PRO 140). Subjects who had undefined or missing data from baseline were excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
days | 286 (0)

6. Secondary Outcome: The Change From Baseline in Circulating Tumor Cells (CTC) Level in the Peripheral Blood.
Description: Reported unit of measure will be the number of CTCs/milliliters. CTCs enumeration will be performed at baseline and at the time of response assessment. Fraction of baseline positive and change from ≥5 CTCs will be recorded and reported.
Time Frame: From date of first treatment until the date of first documented progression or date of death from any cause, whichever came first. From the time of first treatment (T1) until the last study visits completion (up to approximately 16 months).
Population: as for outcome 4
Measure: Number; unit: CTCs/milliliters
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 1
CTCs/milliliters | 22

7. Secondary Outcome: Overall Survival Defined as Time in Months From the Date of First Study Treatment to the Date of Death
Description: Overall survival defined as time in months from the date of first study treatment to the date of death. Patients will be followed from the start of treatment (first dose) until long-term follow up date (up to 2 years post-treatment or death), whichever occurs first, and average survival time will be measured.
Time Frame: Overall survival is calculated by long-term follow-up date - PRO 140 (leronlimab) start date, up to approximately 57 months.
Population: The population consists of all subjects who received at least one dose of leronlimab (PRO 140). Censor subjects are all subjects who had a long-term follow up date.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Leronlimab 525mg
Number analyzed (Participants) | 16
months | 53.60 (3.956)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported from the time of the first treatment and continued up until the final study visit (EOT visit) to evaluate safety of leronlimab (PRO 140) (up to approximately 16 months). All-cause mortality was assessed from first dose through the long-term follow-up period (up to approximately 57 months).
Description: Adverse events were elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the investigator believed were clinically significant to the research subject were reported as adverse events.
Arm/Group | Leronlimab 525mg
All-Cause Mortality (participants affected / at risk) | 12/16
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab 525mg (N=16)
Sepsis (Infections and infestations) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab 525mg (N=16)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Injection site rash (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Localized infection (Infections and infestations) | 1 (2)
Lymphoedema (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Vaccination site reaction (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04504942/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04504942/SAP_002.pdf